CLINICAL TRIAL: NCT05391321
Title: Identification of the Most Suitable Questionnaire to Assess the Sexual Function of Women Living in France After Colorectal Cancer Surgery
Acronym: EVAS-CCR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Limoges (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 87RI21_0062
Record Dates: First submitted 2022-05-20; First posted 2022-05-25 (Actual); Last update posted 2023-12-12 (Actual); Status verified 2023-06

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Intervention Model Description: women will have to answer the 4 sexual quality of life questionnaires. the order of the 4 questionnaires will be randomized
Masking Description: The order of the questionnaires tested will be randomized in each bundle according to the random method. Each bundle will receive a randomization number which will not be known to the patient or the principal investigator.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- administration of quality of sexual life questionnaires (Experimental)
  Interventions: Other: administration of the 4 quality of sexual life questionnaires

INTERVENTIONS:
Other: administration of the 4 quality of sexual life questionnaires — administration of the 4 quality of sexual life questionnaires

SUMMARY:
Sexual quality of life is rarely mentioned by physicians during follow-up consultations, even though it is the source of a significant deterioration in quality of life (QOL).

The assessment of female sexual function is based on self-administered questionnaires. Four questionnaires have been translated and validated in French: FSFI, PISQ-IR, PISQ-12, BISF.

The objective of this project is to determine which questionnaire is acceptable and adapted to a cohort of women living in France who have undergone treatment for rectal cancer

DETAILED DESCRIPTION:
Quality of life (QoL) is often impaired in the aftermath of rectal cancer management due to impaired rectal function and the impact of surgery and radiation therapy on pelvic innervation and the genitourinary sphere. Female sexual function is rarely mentioned by caregivers during follow-up consultations, even though it is a source of significant alteration in the quality of life. Assessment of sexual function is based on self-assessment questionnaires. Most of them were written in English and correspond to the Anglo-Saxon culture. Four questionnaires were translated and validated in French: FSFI, PISQ-IR, PISQ-12, BISF. Two are general sexual HRQOL questionnaires, 2 are sexual HRQOL questionnaires developed for women with genitourinary prolapse.

The identification of the acceptable questionnaire adapted to women living in France will be done through a randomized double-blind study. The duration of patient participation will be 6 months, corresponding to the period of inclusion, collection of informed consent, sending of the questionnaire bundles and collection of the bundles.

ELIGIBILITY:
Inclusion Criteria:

* female
* over 18 years of age
* who have signed the informed consent to participate in the study
* having had rectal or recto-sigmoid cancer at least one year before, whatever the stage, treated by rectal or recto-sigmoid resection with sphincter preservation
* in the course of an eventual adjuvant treatment (chemotherapy or radiotherapy)
* affiliated to the social security system of the health insurance, whatever the system

Exclusion Criteria:

* colon cancer
* pelvic radiotherapy for a pathology other than colorectal cancer
* rectal resection without restoration of continuity (Hartmann or abdominal-perineal amputation)
* peritoneal carcinosis
* colorectal resection for benign lesion
* Inflammatory bowel disease (IBD)
* emergency surgery

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 50 (Estimated)
Dates: Start 2023-05-12 (Actual); Primary Completion 2024-11 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Preference ranking of 4 validated sexual QOL questionnaires in French, FSFI, PISQ-IR, PISQ-12, BISF assessed on the collection of questionnaire returns by patients | 6 months
  Preference ranking of 4 validated sexual QOL questionnaires in French, FSFI, PISQ-IR, PISQ-12, BISF assessed on the collection of questionnaire returns by patients

CONTACTS AND LOCATIONS:
Locations (1):
- Limoges University Hospital, Limoges, France

IPD SHARING:
Plan to Share IPD: No